CLINICAL TRIAL: NCT04915027
Title: Rehabkompassen® - a Novel Digital Tool for Facilitating Patient-tailored Rehabilitation in the Post-acute Continuum of Care After Stroke - A Multicenter Pragmatic Randomized Controlled Trial
Brief Title: Rehabkompassen® - a Patient-centered Digital Follow-up Tool in the Post-stroke Continuum of Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: The Swedish Research Council (Other Government); Forte: Swedish research council for health, working life and welfare (Unknown); Swedish Heart Lung Foundation (Other); Vinnova (Other Government); Strokeförbundet (Unknown); Västerbotten County Council, Sweden (Other Government); Göteborg University (Other); Vastra Gotaland Region (Other Government); Uppsala University (Other); Uppsala County Council, Sweden (Other Government); Karolinska Institutet (Other); Region Stockholm (Other Government); Västmanland County Council, Sweden (Other Government); Värmland County Council, Sweden (Other Government); Sormland County Council, Sweden (Other); Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rehabkompassen®
Record Dates: First submitted 2020-11-11; First posted 2021-06-07 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Stroke
Keywords: Stroke rehabilitation; Patient-tailored rehabilitation; Improvement of daily and social activity; Quality of life; Health economy; Pragmatic randomized clinical trial
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: A pragmatic RCT with allocation ratio 1:1. The permuted block randomization with stratification at each clinic will be used, with random block sizes between 2-8 to ensure participants randomly assigned to intervention respectively control group. All study participants will be followed-up at two occations, at 3- and 12-months after stroke onset. The patients will be identified by participating outpatient clinics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention i.e. with Rehabkompassen® (Experimental): The participants will use the digital graphic Rehabkompassen® at follow-up.
  Interventions: Other: a usual follow-up with Rehabkompassen®
- Control exposure i.e. without Rehabkompassen® (Active Comparator): The participants will use Post-Stroke Checklist at follow-up as recommended by "Socialstyrelsen".
  Interventions: Other: a usual follow-up with Post-Stroke Checklist, i.e. without Rehabkompassen®

INTERVENTIONS:
Other: a usual follow-up with Rehabkompassen® — Rehabkompassen® is a patient-centered digital graphic tool for capturing the patient's rehabilitation needs in the follow-up after stroke.
  Arms: Intervention i.e. with Rehabkompassen®
Other: a usual follow-up with Post-Stroke Checklist, i.e. without Rehabkompassen® — Post-Stroke Checklist consists of eleven questions concerning common and treatable post-stroke problems affecting quality of life.
  Arms: Control exposure i.e. without Rehabkompassen®

SUMMARY:
Stroke is a leading cause of disability and with a heavy burden for the society. Despite the demands from 'Socialstyrelsen' of improving post-acute care, an effective structured follow-up to promote a patient-tailored rehabilitation remains largely lacking in the current stroke care.

The overall aim of this study is to find a cost-effective solution to facilitate patient-tailored rehabilitation that improves daily and social activities and health-related quality of life for persons discharged from the acute care after stroke. We have recently developed a novel digital graphic tool, Rehabkompassen®, which based on patient-reported outcome measurements captures the patient's complex health status after stroke.

Here, this tool will be used in a parallel, open-label, 2-arm prospective and multicenter pragmatic randomized controlled trial between 2022-2026. All participants (n = 1106) will be randomized according to permuted block design; and receive a usual care without (control group, n = 553) or with (intervention group, n = 553) Rehabkompassen®, within 3-month after stroke. The effectiveness of the tool on daily and social activities, quality of life and its health-economic effects will be compared at 12-month follow-up post stroke.

We hypothesize that the digital tool Rehabkompassen® will provide a patient-tailored rehabilitation that improves recovery, independence, and quality of life among people with stroke in a cost-effective way.

DETAILED DESCRIPTION:
Primary research question Does the incorporation of the digital Rehabkompassen® tool in usual care within 3 months after stroke onset result in improved daily and social activities for patients at the 12-month follow-up after stroke onset compared to those receiving usual care with the Post-Stroke Checklist (PSC)?

Secondary research questions

The aim is to investigate the following by comparing usual care with the PSC ® (control group) to usual care with the usage of the digital Rehabkompassen® tool:

1. The improvement of technical and methodological aspects of Rehabkompassen® based on feedback from end-users, including both patients and health care practitioners.
2. The provision of information that affects and/or facilitates the implementation of the Rehabkompassen® tool.
3. The facilitation of triage, clinical assessments, decision-making, the development of a rehabilitation plan, referrals, and outcome evaluations for health care professionals.
4. The influence on secondary outcome measures, including fatigue, depression, anxiety, and other stroke impacts, at the 12-month poststroke follow-up.
5. The impact on patients' health-related quality of life at the 12-month follow-up after stroke onset
6. The demonstration of the cost-effectiveness of the tool.

Study design and patient selection.

In the pilot study

A total of 30 patients will be randomized 1:1 to the intervention group (a usual out-patient visit Rehabkompassen®) or the control group (a usual out-patient visit without Rehabkompassen®) with otherwise identical procedure as that described in the formal RCT below. The aim of the pilot study is to collect information on feasibility of the instrument, key metrics for the formal RCT; and to obtain preliminary efficacy data.

In the formal RCT

All patients who meet the selection criteria, together with the appointment for a usual out-patient follow-up or in the beginning of the inpatient care, receive an invitation to the study. Patients who give their consent are contacted via telephone or in-person by research staff at the local clinic in order to provide oral information about the study. All study participants will be followed-up at 3- and 12-months after stroke onset.

Patients in both control- and intervention groups then receive a message in their inbox at 1177.se. At home or in the inpatient care, patient-participants will be able to fill in the surveys concerning their health by clicking on the links in their e-mail inbox at 1177.se. In an out-patient setting, the questionnaires must be answered no later than one week before the visit. In the inpatient care, patient-participants need to answer the questionnaires in the beginning of the care. In order to facilitate the usage of the digital Rehabkompassen®, research staff will offer technical support via telephone or in-person.

Within 3-month follow-up (Control and Intervention)

A usual care consists of patient's history of disease taken, examination and rehabilitation treatment plan in either inpatient or outpatient settings.

Control group: a usual care + questionnaires

To collect the baseline data, the patient-participants in the control group will fill in only questionnaires of smRSq, SIS-D8 and EQ-5D-5L via 1177.se prior to a usual out-patient follow-up or in the beginning of the inpatient care. The Post-stroke Checklist (PSC) will be used together with the usual care.

Intervention group: a usual care + Rehabkompassen®

The patient-participants will fill in the Rehabkompassen® questionnaires 12. The Rehabkompassen® questionnaires consist of smRSq, SIS, EAT-10, FAS, HAD and EQ-5D-5L. The patient's own graphic Rehabkompassen® will be utilized at the usual care with otherwise identical procedures as the control group.

The replies from the questionnaires (control group) or Rehabkompassen® (intervention group) will be used by doctors / healthcare personnel before the usual in- or out-patient follow-up / team assessment as a basis for triage, and during the usual in- or out-patient follow-up / team assessment as a basis for assessing the patient's rehabilitation needs.

At 12-month follow-up

All participants from control- and intervention group will fill in the Rehabkompassen® questionnaires via 1177.se at home one week prior an out-patient visit. The patient's own graphic Rehabkompassen® will be utilized at the usual out-patient follow-up.

In the primary care study

A total of 30 patients will be randomized 1:1 to the intervention group (a usual out-patient visit Rehabkompassen®) or the control group (a usual out-patient visit without Rehabkompassen®) with similar procedure as that described in the formal RCT above. Compared to the formal RCT, the difference in the primary care study is the first clinical visit will be after 3-month post-stroke and the follow-up visit will be at 6-months after the first clinical visit. The aim of the primary care study is to the feasibility of Rehabkompassen® in the primary care in both qualitative and quantitative ways.

Post-acute continuum of care

In order to understand more about patients experiences regarding the use of the Rehabkompassen®, the qualitative interviews will be conducted within 2 weeks after 12-month follow-up. Meanwhile, the interviews with medical staff will be conducted during the patient recruitment phase to seek the knowledge about their work experience with the tool and their expectation of using the Rehabkompassen® in the post-acute continuum of care.

Technical support and development

Technical support during the study will be carried out by our technical competencies within the research team. The feedback from the end-users (both patient and medical staff) at the 3-month follow-up and during the whole using process will be used to further develop and refine the tool by our technical competencies within the research team.

Study Design, Randomization and blinding

To evaluate the hypotheses in this proposed study, we have designed a parallel, open-label, 2-arm prospective multicenter pragmatic RCT with allocation ratio 1:1. We intend to use permuted block randomization with stratification at each clinic. We will use random block sizes between 2-8 to ensure participants randomly assigned to intervention respectively control group 15. The randomization list will be created centrally by REDCap, and handled by an investigator who will not be involved in outcome assessment or the patient's treatment.

Patients will be identified by approximately 15 participating centers from at least 4 regions. In a three-year recruitment period, we have estimated that approximately 21 000 stroke patients need structured follow-up in the catchment area. All patient-participants will receive two follow-ups, i.e one within 3-month and another at 12-month after stroke onset.

Estimated sample size and power

The study is dimensioned to reach 90% in the analysis of the two primary outcomes at a significance level of 2.5% for each individual test, to account for planned correction for multiple comparison with a target familywise error rate of 5%.

Sample size calculations have been performed assuming a difference of 4 points in SIS-p between, which is well below any concluded smallest important differences reported in the literature 20. A power analysis has been conducted using Monte Carlo simulations, in which SIS-p data for the control group was generated from a beta distribution with parameters α = 1.1 and β = 0.5, while Rehabkompassen® was generated under the assumption of α = 1.1 and β = 0.385. This corresponds to approximately to a mean value of 70 and standard deviation of 28 for the control group, in line with what Guidetti et al 18 reported for population of stroke patients at 12 months after stroke, and a difference of 4 points in mean values between groups. Under these assumptions, results showed that we need to include 940 patients to detect a statistically significant difference for SIS-p using a proportional odds model. The setting of the simulation corresponds to an odds ratio between groups of 1.5.

The marginal distribution of mRS score used for dimensioning was based on aggregated unpublished data from the Swedish Stroke Register (Riksstroke), collected 12-month after a stroke among Swedish patients: 0: 22.4%, 1: 18.0%, 2: 18.0 %, 3: 16.8%, 4: 11.1%, 5: 4.3%, 6: 9.4%. A sample size of 940 patients (470 in each group) is sufficient to detect a true odds ratio of 0.67 using an ordinal proportional odds model. The function popower from the package Hmisc in the statistical software R was used in this calculation.

Thus, 940 patients are required for both primary outcomes. To account for a 15% rate of patients being lost to follow up, we plan to recruit 1106 patients to the study.

Analysis and statistics

Statistical methods for primary and secondary outcomes Group differences in the mRS and SIS-p scores at the 12-month follow-up will be tested using ordinal logistic (proportional odds) regression, adjusted for site with fixed effects. For the SIS-p score, models will also be adjusted for the baseline SIS-p score, with natural cubic splines to account for nonlinearity in the association. The results from the analyses will be presented as odds ratios with corresponding 95% confidence intervals and p values.

For the two primary outcomes, adjustments of the significance levels of the individual tests will be performed using the Holm-Bonferroni method to ensure that the familywise error rate will not be inflated above 0.05.

Secondary outcomes on an ordinal scale will be analysed similarly using ordinal logistic regression. All analyses will primarily be conducted in accordance with the intention-to-treat principle. As complementary analyses, per-protocol analyses will be performed using data from patients with full availability of primary variables and predefined criteria for adherence. Further details about the statistical analyses will be predefined and published in a separate statistical analysis plan. A data management plan has been established, providing details of the handling, organization and storage of study data.

A statistical significance level of p < 0.05 (two-tailed) will be applied to all analyses. For the two primary outcomes, adjustments of the significance levels of the individual tests will be performed using the Holm-Bonferroni method to ensure that the familywise error rate will not be inflated above 0.05.

Methods for additional analyses (e.g., subgroup analyses) Subgroup analyses, e.g., based on age (< 65 years, 65-80 years and > 80 years), sex (male and female), stroke severity (NIHSS score; mild, 0-8 moderate, 9-15 and severe, > 15), stroke type (ischaemic vs. haemorrhagic), treatment with tissue plasminogen activator and/or thrombectomy (yes or no), and geographical region, will be conducted as complementary analyses.

Methods in analysis to handle protocol nonadherence and any statistical methods to handle missing data All analyses will be conducted in accordance with the intention-to-treat principle. Multiple imputation of missing data will be employed in the primary analysis using multiple imputation by chained equation (MICE). As sensitivity analyses, per-protocol analyses will be performed using data from patients with fully available data for the primary variables and no protocol violations. The per-protocol dataset will be predefined in the statistical analysis plan of the study.

Time plan and implementation

The proposed study has already started the recruitment phase as from the beginning of 2022, aiming to recruit 15% of the participants this year. Approximately 40% and 45% of the sample size will be recruited in year 2023 and 2024 respectively. The 12-month follow-up will be completed at the end of 2027 followed by data analysis, manuscript preparations and submissions in 2027 and afterwards.

ELIGIBILITY:
Inclusion criteria are

1. Adults aged 18 years or older.
2. With a stroke diagnosis

Time since stroke onset:

3a) For the big RCT group, Individuals must be within the first 4 months after stroke, starting from Day 1 after the occurrence of the stroke.

3b) For primary care group, Individuals 3 months after stroke

Exclusion criteria are

1. Unable to answer the evaluation questions.
2. Unable to see the Rehabkompassen®graph.
3. Not using BankID, an e-identification tool commonly used in Sweden.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1106 (Estimated)
Dates: Start 2020-08-26 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Daily activities | 12 months follow-up after stroke
  The simplified modified Rankin Scale questionnaire (smRSq) will be used to measure daily activities and functional status. The smRSq is based on the yes/no responses to five questions, which in turn results an ordinal data of seven categories (0-6) of the modified Rankin Scale. A favorable outcome will be defined as mRS score of 0-2 (no symptoms to independent but with minor disability). A poor outcome will be defined as mRS score of 3-5 (disability but able to walk to bed-bound and in need of full nursing care) or 6 (death).
Social activities | 12 months follow-up after stroke
  Stroke Impact Scale 3.0 (SIS)-participation (SIS-p) will be used to measure social activities. SIS-p is the dominant problem among persons after stroke reported in previous Swedish stroke RCTs; but not covered by smRSq. The SIS-p score ranges from 0-100 and the higher the score the less impact of stroke.

SECONDARY OUTCOMES:
Health-related quality of life | 12 months follow-up after stroke
  Health-related quality of life will be measured by five-level EuroQoL 5-dimension (EQ- 5D-5L) at both follow-ups in all participants. EQ-5D is a validated instrument that has often been used in RCTs. It consists of two parts: a visual analogue scale and a descriptive system covering five dimensions of health (mobility, hygiene, usual activities, pain/discomfort, and anxiety/depression) with five response alternatives (ranging from no problems to extreme problems). The latter can be translated to index value with anchor points 0 (death) and 1 (full health), which corresponds to a QALY score.
Stroke impacts | 12 months follow-up after stroke
  Stroke impacts will be assessed by the Stroke Impact Scale 3.0 (SIS) except the participation domain. SIS is a patient-reported, stroke-specific, outcome measurement containing 59 questions with eight domains, namely strength, memory/ cognition, feelings/ emotions, communication, personal activities of daily living (ADL), instrumental ADL, mobility, and motor impact. Each question is answered using the Likert scale ranging from 1 to 5 with higher scores indicating better outcomes. Also, the SIS includes a visual analogue scale where 0 represents no perceived stroke recovery and 100 represents full recovery.
Health-economic evaluation | 12 months follow-up after stroke
  The cost-effectiveness will be assessed in term of the quality-adjusted life year (QALY), that will be calculated by the utilities multiplying the time spent in each health state.
Clinicians' usability | 3 months follow-up after stroke
  System usability scale consists of a 10-item questionnaire with five response options for respondents from strongly agree to strongly disagree.
End-users' experiences and feedback | 3 months follow-up after stroke
  End-users' satisfaction questionnaire consists of a 17-item questionnaire concerning their experiences of using the Rehabkompassen®. Each question is answered using the Likert scale ranging from 1 to 5 with higher scores indicating better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolei Hu, MD PhD, Principal Investigator — Umeå University
Locations (1):
- Umeå University Hospital, Umeå, Sweden

REFERENCES:
- [Background] Hu X, Wester P, Stibrant Sunnerhaagen K. [Evidence-based methods in the clinical practice in updated Swedish national stroke guidelines]. Lakartidningen. 2018 Dec 17;115:FDIX. Swedish. PMID 30561751
- [Background] Hudon C, Fortin M, Haggerty JL, Lambert M, Poitras ME. Measuring patients' perceptions of patient-centered care: a systematic review of tools for family medicine. Ann Fam Med. 2011 Mar-Apr;9(2):155-64. doi: 10.1370/afm.1226. PMID 21403143
- [Background] Magaard G, Wester P, Levi R, Lindvall P, Gustafsson E, Nazemroaya Sedeh A, Lonnqvist M, Berggren S, Nyman K, Hu X. Identifying Unmet Rehabilitation Needs in Patients After Stroke With a Graphic Rehab-CompassTM. J Stroke Cerebrovasc Dis. 2018 Nov;27(11):3224-3235. doi: 10.1016/j.jstrokecerebrovasdis.2018.07.013. Epub 2018 Aug 8. PMID 30097401
- [Background] Devlin NJ, Brooks R. EQ-5D and the EuroQol Group: Past, Present and Future. Appl Health Econ Health Policy. 2017 Apr;15(2):127-137. doi: 10.1007/s40258-017-0310-5. PMID 28194657
- [Background] Copas AJ, Lewis JJ, Thompson JA, Davey C, Baio G, Hargreaves JR. Designing a stepped wedge trial: three main designs, carry-over effects and randomisation approaches. Trials. 2015 Aug 17;16:352. doi: 10.1186/s13063-015-0842-7. PMID 26279154
- [Background] Hargreaves JR, Copas AJ, Beard E, Osrin D, Lewis JJ, Davey C, Thompson JA, Baio G, Fielding KL, Prost A. Five questions to consider before conducting a stepped wedge trial. Trials. 2015 Aug 17;16:350. doi: 10.1186/s13063-015-0841-8. PMID 26279013
- [Background] EFFECTS Trial Collaboration. Safety and efficacy of fluoxetine on functional recovery after acute stroke (EFFECTS): a randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2020 Aug;19(8):661-669. doi: 10.1016/S1474-4422(20)30219-2. PMID 32702335
- [Background] White IR, Horton NJ, Carpenter J, Pocock SJ. Strategy for intention to treat analysis in randomised trials with missing outcome data. BMJ. 2011 Feb 7;342:d40. doi: 10.1136/bmj.d40. PMID 21300711
- [Background] Optimising Analysis of Stroke Trials (OAST) Collaboration; Bath PM, Gray LJ, Collier T, Pocock S, Carpenter J. Can we improve the statistical analysis of stroke trials? Statistical reanalysis of functional outcomes in stroke trials. Stroke. 2007 Jun;38(6):1911-5. doi: 10.1161/STROKEAHA.106.474080. Epub 2007 Apr 26. PMID 17463316
- [Background] Savitz SI, Lew R, Bluhmki E, Hacke W, Fisher M. Shift analysis versus dichotomization of the modified Rankin scale outcome scores in the NINDS and ECASS-II trials. Stroke. 2007 Dec;38(12):3205-12. doi: 10.1161/STROKEAHA.107.489351. Epub 2007 Nov 1. PMID 17975102
- [Background] Hu X, Jonzen K, Karlsson M, Lindahl OA. Assessments of a novel digital follow-up tool Rehabkompassen(R) to identify rehabilitation needs among stroke patients in an outpatient setting. Digit Health. 2022 Jun 3;8:20552076221104662. doi: 10.1177/20552076221104662. eCollection 2022 Jan-Dec. PMID 35677783
- [Background] Hu X, Jonzen K, Lindahl OA, Karlsson M, Norstrom F, Lundstrom E, Sunnerhagen KS. Digital Graphic Follow-up Tool (Rehabkompassen) for Identifying Rehabilitation Needs Among People After Stroke: Randomized Clinical Feasibility Study. JMIR Hum Factors. 2022 Jul 29;9(3):e38704. doi: 10.2196/38704. PMID 35904867
- [Derived] Hu X, Liv P, Lundstrom E, Norstrom F, Lindahl O, Borg K, Sunnerhagen KS. Study protocol for a randomized, controlled, multicentre, pragmatic trial with Rehabkompassen(R)-a digital structured follow-up tool for facilitating patient-tailored rehabilitation in persons after stroke. Trials. 2023 Oct 6;24(1):650. doi: 10.1186/s13063-023-07673-7. PMID 37803460